CLINICAL TRIAL: NCT04782323
Title: A Phase 2, Randomized, Observer-blind, Antigen and Adjuvant Dose Ranging Clinical Study to Evaluate Safety and Immunogenicity of Different Formulations of MF59 Adjuvanted Quadrivalent Subunit Inactivated Cell-derived Influenza Vaccine (aQIVc) in Older Adults ≥50 Years of Age
Brief Title: Safety and Immunogenicity of Different Formulations of an MF59-Adjuvanted Influenza Vaccine in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V201_01
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a parallel-group dose-ranging study with 8 arms that is participant, investigator and observer-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group A aQII-1 Investigational (Experimental)
  Interventions: Drug: aQII-1
- Group B aQII-3 Investigational (Experimental)
  Interventions: Drug: aQII-3 Investigational
- Group C aQII-6 Investigational (Experimental)
  Interventions: Drug: aQII-6 Investigational
- Group D aQII-7 Investigational (Experimental)
  Interventions: Other: aQII-7 Investigational
- Group E aQII-9 Investigational (Experimental)
  Interventions: Drug: aQII-9 Investigational
- Group F aQII-10 Investigational (Experimental)
  Interventions: Drug: aQII-10 Investigational
- Group G aQII-11 Investigational (Experimental)
  Interventions: Drug: aQII-11 Investigational
- Group H Licensed QII Active Comparator (Active Comparator)
  Interventions: Drug: Licensed QII Active Comparator

INTERVENTIONS:
Drug: aQII-1 — Biological/Vaccine: Investigational aQII-1 Investigational MF59 Adjuvanted Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Group A aQII-1 Investigational
Drug: aQII-3 Investigational — Biological/Vaccine: Investigational aQII-3 Investigational MF59 Adjuvanted Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Group B aQII-3 Investigational
Drug: aQII-6 Investigational — Biological/Vaccine: Investigational aQII-6 Investigational MF59 Adjuvanted Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Group C aQII-6 Investigational
Other: aQII-7 Investigational — Biological/Vaccine: Investigational aQII-7 Investigational MF59 Adjuvanted Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Group D aQII-7 Investigational
Drug: aQII-9 Investigational — Biological/Vaccine: Investigational aQII-9 Investigational MF59 Adjuvanted Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Group E aQII-9 Investigational
Drug: aQII-10 Investigational — Biological/Vaccine: Investigational aQII-10 Investigational MF59 Adjuvanted Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Group F aQII-10 Investigational
Drug: aQII-11 Investigational — Biological/Vaccine: Investigational aQII-11 Investigational MF59 Adjuvanted Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Group G aQII-11 Investigational
Drug: Licensed QII Active Comparator — Biological/Vaccine: Licensed QII Licensed Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Group H Licensed QII Active Comparator

SUMMARY:
This Phase 2, randomized, observer-blind, antigen and adjuvant dose-ranging Clinical study is evaluating different formulations of MF59-Adjuvanted Quadrivalent Subunit Inactivated Influenza Vaccine. Approximately 800 subjects are to be randomized into 1 of 8 possible treatment groups. Immunogenicity and safety will be assessed in the overall study population (adults ≥50 years and above) and in the age subgroups ≥50-64 years and ≥65 years. Data from this study will be used to select the optimal dose to be tested in the pivotal Phase 3 immunogenicity and safety study in older adults.

Disclosure Statement: This is a parallel-group dose-ranging study with 8 arms that is participant, investigator and observer-blinded.

ELIGIBILITY:
INCLUSION CRITERIA:

In order to participate in this study, all subjects must meet ALL of the inclusion criteria described.

1. Individuals ≥50 years of age on the day of informed consent.
2. Individuals who have voluntarily given written consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
3. Individuals who can comply with study procedures including follow-up .
4. Males, females of non-childbearing potential or females of childbearing potential who are using an effective birth control method, at least 30 days prior to informed consent, which they intend to use for at least 2 months after the study vaccination.

EXCLUSION CRITERIA:

In order to participate in this study, all subjects must not meet ANY of the exclusion criteria described below:

1. Females of childbearing potential who are pregnant, lactating, or who have not adhered to a specified set of contraceptive methods from at least 30 days prior to informed consent and who do not plan to do so for at least 2 months after the study vaccination.
2. Progressive, unstable or uncontrolled clinical conditions.
3. Hypersensitivity, including allergy, to any component of vaccines whose use is foreseen in this study.
4. History of any medical condition considered an adverse event of special interest (AESI).
5. Known history of Guillain-Barré syndrome or another demyelinating disease such as encephalomyelitis and transverse myelitis.
6. Clinical conditions representing a contraindication to intramuscular administration of vaccines or blood draw.
7. Abnormal function of the immune system resulting from:

   1. Clinical conditions.
   2. Systemic administration of corticosteroids (PO/IV/IM) at a dose of ≥20 mg/day of prednisone or equivalent for more than 14 consecutive days within 90 days prior to informed consent.
   3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
8. Receipt of immunoglobulins or any blood products within 180 days prior to informed consent.
9. Receipt of an investigational or non-registered medicinal product within 30 days prior to vaccination.
10. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine within 28 days from the study vaccines.
11. Study personnel or immediate family or household member of study personnel.
12. Receipt of any influenza vaccine within 6 months prior to vaccination in this study, or plan to receive an influenza vaccine during the study period.
13. Acute (severe) febrile illness.
14. Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Therapeutic Area Head, Study Chair — Seqirus
Locations (30):
- Australia (11):
  - 03607 - PCRN_Paratus Clinical Research, Bruce, Australian Capital Territory
  - 03605 - PCRN_Paratus Clinical Research (Central Coast), Blacktown, New South Wales
  - 3610- Emeritis Research, Botany, New South Wales
  - 3609 - Northern Beaches Clinical Research [NSW], Brookvale, New South Wales
  - 03602 - PCRN_Paratus Clinical Research,(Western Sydney) [NSW], Kanwal, New South Wales
  - 03608 - Australian Clinical Research Network - ACRN [NSW], Maroubra, New South Wales
  - 03604 - University of the Sunshine Coast Clinical Trials Centre, Morayfield, Queensland
  - 03603 - University of the Sunshine Coast, Sippy Downs, Queensland
  - 03601 - AusTrials Taringa [QLD], Taringa, Queensland
  - 03606 - AusTrials Tarragindi (Aus Trial Wellers Hill)[QLD], Tarragindi, Queensland
  - 3611 - The University of Melbourne Peter Doherty Institute for Infection and Immunity, Melbourne, Victoria
- New Zealand (6):
  - 55402- PCRN_Southern Clinical Trials Waitemata, Birkenhead, Auckland
  - 55401- PCRN_Southern Clinical Trials Totara, New Lynn, Auckland
  - 55406 - Optimal Clinical Trials, Auckland
  - 55404- PCRN_Southern Clinical Trials Christchurch, Christchurch
  - 55403-PCRN_Lakeland Clinical Trials Waikato, Hamilton
  - 55405 - PCRN_Lakeland Clinical Trials, Rotorua
- Philippines (5):
  - 60801 - De La Salle Medical and Health Sciences Institute, Dasmariñas, Cavite
  - 60802 - West Visayas University Medical Center, Jaro, Iloilo City
  - 60805 - Manila Doctors' Hospital, Ermita, Manila
  - 60804 - Quirino Memorial Medical Center, Quezon City, Quezon
  - 60803 - Philippine General Hospital, Manila
- South Africa (8):
  - 71003- Newtown Clinical Research, Newtown, Johannesburg
  - 71005 South Africa Haylene71005 - Tiervlei Trial Centre -- Karl Bremer Hospital, Bellville
  - 71002 - JOSHA Research, Bloemfontein
  - 71011 - Farmovs, Bloemfontein
  - 71004 - Tread Research -- Tygerberg Hospital, Cape Town
  - 71006 - Mzansi Ethical Research Centre (MERC), Mpumalanga
  - 71009 - Be Part Yoluntu Centre, Paarl
  - 71001 - Wits Clinical Researc - Chris Hani Baragwanath Academic Hospital, Soweto

IPD SHARING:
Plan to Share IPD: Yes
SEQIRUS supports the release of anonymized subject-level and study-level data in compliance with regulatory requirements, including Clinical Documents which are part of the CTD modules submitted to regulatory agencies for public release.
  Summary results disclosure is either in document form (e.g., ICH E3 Clinical Study Report synopsis) or structured data form (such as summary results in ClinicalTrials.gov (United States) or eudract.ema.europa.eu (EU Clinical Trial Registry [EU CTR])
Supporting Information: Study Protocol, SAP
Time Frame: Time Frame:
  SEQIRUS discloses results from clinical studies within 12 months of last patient last visit (LPLV) unless otherwise mandated by local laws or regulations.
Access Criteria: SEQIRUS will consider requests from qualified scientific and medical researchers to disclose protocols, anonymized subject-level data and study-level data when there is medical, scientific and/or public health interest to ensure the safe use of a Seqirus product licensed on or after 1 January 2014 in the United States (US) and/or the European Union (EU). This applies to Seqirus-sponsored interventional studies initiated after 27 September 2007 and ongoing as of 26 December 2007, that have been included as part of a US or EU submission package which received approval in US and EU on or after 1 January 2014 and have been accepted for publication
URL: https://www.seqirus.us/partnering

RESULTS

PARTICIPANT FLOW:
Groups:
- Group H Licensed QII Active Comparator: Licensed QII Active Comparator: Biological/Vaccine: Licensed QII Active Comparator Licensed Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
Period: Overall Study
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Started | 98 | 107 | 107 | 103 | 106 | 108 | 101 | 109
Completed | 96 | 106 | 105 | 103 | 105 | 105 | 99 | 106
Not Completed | 2 | 1 | 2 | 0 | 1 | 3 | 2 | 3
Not completed — Death | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2
Not completed — randomization in error | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational | Total
Number analyzed (Participants) | 98 | 107 | 107 | 103 | 106 | 108 | 101 | 109 | 839
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 55 | 53 | 52 | 58 | 58 | 54 | 60 | 442
  >=65 years | 46 | 52 | 54 | 51 | 48 | 50 | 47 | 49 | 397
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.68) | 63.6 (8.91) | 63.6 (8.1) | 63.3 (8.48) | 62.8 (8.22) | 63.5 (8.82) | 64.4 (9.12) | 63.1 (8.5) | 63.5 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 62 | 63 | 63 | 57 | 49 | 53 | 59 | 475
  Male | 29 | 45 | 44 | 40 | 49 | 59 | 48 | 50 | 364
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 56 | 66 | 51 | 56 | 61 | 58 | 58 | 63 | 469
  black or african american | 11 | 16 | 15 | 11 | 15 | 13 | 13 | 17 | 111
  asian | 21 | 14 | 22 | 20 | 18 | 18 | 16 | 18 | 147
  native hawaiian or other pacific islander | 0 | 2 | 3 | 3 | 0 | 2 | 4 | 1 | 15
  other | 10 | 9 | 16 | 13 | 12 | 17 | 10 | 10 | 97
Region of Enrollment [Number; unit: participants]
  New Zealand | 29 | 32 | 32 | 30 | 30 | 33 | 29 | 31 | 246
  Philippines | 15 | 11 | 16 | 17 | 12 | 13 | 12 | 13 | 109
  South Africa | 18 | 27 | 21 | 20 | 26 | 24 | 20 | 25 | 181
  Australia | 36 | 37 | 38 | 36 | 38 | 38 | 40 | 40 | 303
vaccinated within 3 previous influenza season [Count of Participants; unit: Participants]
  Yes | 60 | 66 | 61 | 68 | 62 | 65 | 61 | 63 | 506
  No | 38 | 41 | 46 | 35 | 44 | 43 | 40 | 46 | 333

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) for the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Hemagglutination Inhibition (HI) Assay and for A/H3N2 Strain Using Microneutralization Assay
Time Frame: [28 days post-vaccination]
Population: Per Protocol Set (PPS) Immunogenicity: All subjects in the FAS Immunogenicity who
  * Correctly received the vaccine (ie, received the vaccine to which the subject was randomized within the defined window).
  * Had no CSR-reportable PD leading to exclusion (ie, impacting the results) as defined prior to unblinding.
  * Had immunogenicity assessments within the window of -7/+21 days around the Day 29 visit, and Day 1 sample taken.
  * Were not excluded due to other reason defined prior to unblinding.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 95 | 105 | 106 | 99 | 102 | 104 | 95 | 104
titer
  A/H1N1 Day 1 HI GMT | 42.31 [34.3 to 52.2] | 40.39 [33.1 to 49.3] | 48.29 [39.6 to 58.9] | 49.31 [40.1 to 60.6] | 46.19 [37.7 to 56.6] | 47.50 [38.9 to 58.1] | 46.92 [38.0 to 57.9] | 37.24 [30.5 to 45.5]
  A/H1N1 Day 29 HI GMT | 228.11 [181.2 to 287.1] | 175.95 [141.3 to 219.1] | 200.22 [161.1 to 248.8] | 225.66 [180.0 to 282.8] | 223.37 [179.0 to 278.8] | 243.16 [195.2 to 302.9] | 270.55 [215.0 to 340.5] | 220.29 [176.8 to 274.5]
  B/Yamagata Day 1 HI GMT | 15.02 [12.5 to 18.0] | 16.7 [14.1 to 19.8] | 20.83 [17.6 to 24.7] | 18.35 [15.4 to 21.9] | 15.51 [13.0 to 18.5] | 16.41 [13.8 to 19.5] | 17.13 [14.3 to 20.5] | 16.00 [13.5 to 19.0]
  B/Yamagata Day 29 HI GMT | 47.73 [40.0 to 56.9] | 47.46 [40.2 to 56.1] | 59.74 [50.6 to 70.5] | 62.34 [52.5 to 74.1] | 61.36 [51.8 to 72.7] | 63.21 [53.5 to 74.7] | 68.14 [57.2 to 81.2] | 69.13 [58.5 to 81.7]
  B/Victoria Day 1 HI GMT | 58.85 [48.0 to 72.1] | 74.31 [61.2 to 90.1] | 65.27 [53.9 to 79.1] | 68.00 [55.7 to 83.0] | 62.26 [51.2 to 75.7] | 63.72 [52.5 to 77.4] | 79.15 [64.6 to 97.0] | 64.13 [52.8 to 77.8]
  B/Victoria Day 29 HI GMT | 145.12 [124.5 to 169.1] | 146.85 [126.9 to 169.9] | 138.29 [119.7 to 159.8] | 141.84 [122.1 to 164.8] | 178.15 [153.7 to 206.4] | 160.54 [138.7 to 185.8] | 181.93 [156.1 to 212.0] | 186.06 [160.8 to 215.3]
  A/H3N2 Day 1 MN GMT | 35.31 [29.2 to 42.7] | 31.61 [26.4 to 37.8] | 32.05 [26.8 to 38.3] | 32.48 [27.0 to 39.1] | 36.83 [30.7 to 44.2] | 32.71 [27.3 to 39.2] | 30.80 [25.5 to 37.2] | 27.15 [22.7 to 32.5]
  A/H3N2 Day 29 MN GMT | 146.59 [124.0 to 173.3] | 142.04 [121.2 to 166.5] | 178.87 [152.8 to 209.4] | 185.07 [157.1 to 218.0] | 193.02 [164.3 to 226.8] | 189.17 [161.3 to 221.9] | 197.27 [166.9 to 233.1] | 157.90 [134.6 to 185.3]

2. Primary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) (GMR is GMT Ratio of aQII Formulation/Licensed QII) for the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by HI Assay and for A/H3N2 Strain Using MN Assay
Time Frame: 28 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 105 | 106 | 99 | 102 | 104 | 95 | 104
Ratio
  A/H1N1 HI GMR (aQII/QII) | 0.77 [0.56 to 1.06] | 0.88 [0.64 to 1.20] | 0.99 [0.72 to 1.36] | 0.98 [0.71 to 1.35] | 1.07 [0.78 to 1.46] | 1.19 [0.86 to 1.64] | 0.97 [0.70 to 1.33]
  B/Yamagata HI GMR (aQII/QII) | 0.99 [0.78 to 1.27] | 1.25 [0.98 to 1.59] | 1.31 [1.02 to 1.67] | 1.29 [1.01 to 1.64] | 1.32 [1.04 to 1.69] | 1.43 [1.12 to 1.83] | 1.45 [1.14 to 1.84]
  B/Victoria HI GMR (aQII/QII) | 1.01 [0.82 to 1.25] | 0.95 [0.77 to 1.18] | 0.98 [0.79 to 1.21] | 1.23 [0.99 to 1.52] | 1.11 [0.9 to 1.37] | 1.25 [1.01 to 1.56] | 1.28 [1.04 to 1.58]
  A/H3N2 MN GMR (aQII/QII) | 0.97 [0.77 to 1.22] | 1.22 [0.97 to 1.53] | 1.26 [1.00 to 1.59] | 1.32 [1.04 to 1.66] | 1.29 [1.03 to 1.62] | 1.35 [1.06 to 1.70] | 1.08 [0.86 to 1.36]

3. Primary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving Seroconversion for the A/H1N1, B/Victoria and B/Yamagata Strains by HI Assay and A/H3N2 Strain Using MN Assay
Description: Seroconversion is defined as ≥4-fold increase in titer postvaccination in those with pre-vaccination titer above or equal to the Lower Limit of Quantitation (LLOQ) (≥1:10), or a post-vaccination titer ≥1:40 for subjects with baseline titer below the LLOQ (1:10) for HI titers
Time Frame: 28 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 95 | 105 | 106 | 99 | 102 | 104 | 95 | 104
percentage of subjects
  A/H1N1 HI seroconversion Day 29 | 55.8 [45.2 to 66.0] | 53.3 [43.3 to 63.1] | 51.9 [42.0 to 61.7] | 54.5 [44.2 to 64.6] | 57.8 [47.7 to 67.6] | 58.7 [48.6 to 68.2] | 60.0 [49.4 to 69.9] | 57.7 [47.6 to 67.3]
  B/Yamagata HI seroconversion Day 29 | 35.8 [26.2 to 46.3] | 35.2 [26.2 to 45.2] | 42.5 [32.9 to 52.4] | 46.5 [36.4 to 56.8] | 41.2 [31.5 to 51.4] | 46.2 [36.3 to 56.2] | 48.4 [38.0 to 58.9] | 51.0 [41.0 to 60.9]
  B/Victoria HI seroconversion Day 29 | 32.6 [23.4 to 43.0] | 25.7 [17.7 to 35.2] | 22.6 [15.1 to 31.8] | 26.3 [17.9 to 36.1] | 35.3 [26.1 to 45.4] | 38.5 [29.1 to 48.5] | 34.7 [25.3 to 45.2] | 34.6 [25.6 to 44.6]
  A/H3N2 MN seroconversion Day 29 | 53.7 [43.2 to 64.0] | 54.3 [44.3 to 64.0] | 67.0 [57.2 to 75.8] | 62.6 [52.3 to 72.1] | 59.8 [49.6 to 69.4] | 62.5 [52.5 to 71.8] | 71.6 [61.4 to 80.4] | 65.4 [55.4 to 74.4]

4. Primary Outcome: Immunogenicity Endpoint: Percentage of Subjects With HI Titer ≥1:40 for A/H1N1, B/Yamagata and B/Victoria Strains (HI Assay)
Time Frame: 28 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 95 | 105 | 106 | 99 | 102 | 104 | 95 | 104
percentage of subjects
  A/H1N1 Day 1 | 66.3 [55.9 to 75.7] | 60.0 [50.0 to 69.4] | 67.9 [58.2 to 76.7] | 71.7 [61.8 to 80.3] | 68.6 [58.7 to 77.5] | 66.3 [56.4 to 75.3] | 66.3 [55.9 to 75.7] | 51.0 [41.0 to 60.9]
  A/H1N1 Day 29 | 95.8 [89.6 to 98.8] | 94.3 [88.0 to 97.9] | 96.2 [90.6 to 99.0] | 93.9 [87.3 to 97.7] | 92.2 [85.1 to 96.6] | 95.2 [89.1 to 98.4] | 98.9 [94.3 to 100.0] | 90.4 [83.0 to 95.3]
  B/Yamagata day 1 | 22.1 [14.2 to 31.8] | 29.5 [21.0 to 39.2] | 34.9 [25.9 to 44.8] | 28.3 [19.7 to 38.2] | 22.5 [14.9 to 31.9] | 25.0 [17.0 to 34.4] | 27.4 [18.7 to 37.5] | 26.9 [18.7 to 36.5]
  B/Yamagata day 29 | 74.7 [64.8 to 83.1] | 68.6 [58.8 to 77.3] | 78.3 [69.2 to 85.7] | 84.8 [76.2 to 91.3] | 77.5 [68.1 to 85.1] | 75.0 [65.6 to 83.0] | 80.0 [70.5 to 87.5] | 79.8 [70.8 to 87.0]
  B/Victoria Day 1 | 72.6 [62.5 to 81.3] | 78.1 [69.0 to 85.6] | 81.1 [72.4 to 88.1] | 79.8 [70.5 to 87.2] | 71.6 [61.8 to 80.1] | 76.0 [66.6 to 83.8] | 78.9 [69.4 to 86.6] | 74.0 [64.5 to 82.1]
  B/Victoria Day 29 | 94.7 [88.1 to 98.3] | 92.4 [85.5 to 96.7] | 95.3 [89.3 to 98.5] | 94.9 [88.6 to 98.3] | 97.1 [91.6 to 99.4] | 97.1 [91.8 to 99.4] | 94.7 [88.1 to 98.3] | 98.1 [93.2 to 99.8]

5. Primary Outcome: Safety Endpoint: Percentage of Subjects With Solicited Local or Systemic Reactions
Description: Percentage of subjects with at least one solicited AE Day 1 through Day 7 after study vaccination
Time Frame: 7 days post-vaccination
Population: Solicited Safety Set, defined as all subjects in the Exposed Set with any solicited AE data.
Measure: Count of Participants; unit: Participants
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 96 | 107 | 107 | 103 | 105 | 105 | 101 | 108
Participants
  solicited AEs | 44 | 69 | 71 | 76 | 85 | 73 | 60 | 82
  Solicited local AEs | 29 | 55 | 63 | 68 | 72 | 57 | 55 | 73
  Solicited systemic AEs | 34 | 48 | 49 | 59 | 66 | 52 | 46 | 64

6. Primary Outcome: Safety Endpoint: The Percentage of Subjects With Any Unsolicited Adverse Events
Description: The percentage of subjects with at least one unsolicited AE from Day 1 to Day 29.
  Related AEs = considered at least possibly related to study vaccination by the investigator
Time Frame: 28 days post-vaccination
Population: Unsolicited Safety Set, defined as all subjects in the Exposed Set with any unsolicited AE data
Measure: Count of Participants; unit: Participants
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 97 | 107 | 108 | 103 | 106 | 107 | 101 | 109
Participants
  Any Unsolicited AE | 29 | 27 | 26 | 30 | 32 | 26 | 30 | 30
  Any Related Unsolicited AE | 9 | 7 | 11 | 14 | 15 | 9 | 6 | 16

7. Primary Outcome: Safety Endpoint: The Percentage of Subjects With Serious Adverse Events (SAEs), AEs Leading to Withdrawal, Adverse Events of Special Interest (AESI) and Medically Attended Adverse Events (MAAEs)
Time Frame: 28 days post-vaccination
Population: Unsolicited Safety Set, defined as all subjects in the Exposed Set with any unsolicited AE data
Measure: Count of Participants; unit: Participants
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 97 | 107 | 108 | 103 | 106 | 107 | 101 | 109
Participants
  Any Serious Unsolicited AE | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Any Unsolicited AE of Special Interest | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Medically Attended AE | 13 | 5 | 5 | 8 | 4 | 9 | 9 | 7
  Any Unsolicited AE Leading to Withdrawal from the Study | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any deaths | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Safety Endpoint: The Percentage of Subjects With Serious Adverse Events (SAEs), AEs Leading to Withdrawal, Adverse Events of Special Interest (AESI) and Medically Attended Adverse Events (MAAEs) During the Entire Study Period
Time Frame: 180 days post-vaccination
Population: Unsolicited Safety Set, defined as all subjects in the Exposed Set with any unsolicited AE data
Measure: Count of Participants; unit: Participants
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 97 | 107 | 108 | 103 | 106 | 107 | 101 | 109
Participants
  Any Serious Unsolicited AE | 8 | 1 | 1 | 3 | 5 | 3 | 2 | 2
  Any Related Serious Unsolicited AE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Any Unsolicited AE of Special Interest | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Any Medically Attended AE | 20 | 15 | 13 | 18 | 14 | 21 | 20 | 16
  Any Unsolicited AE Leading to Withdrawal from the Study | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Deaths | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0

9. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) for the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Microneutralization (MN) Assay
Time Frame: 28 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 95 | 105 | 106 | 99 | 102 | 104 | 95 | 104
titer
  A/H1N1 Day 1 | 44.55 [34.6 to 57.4] | 29.77 [23.4 to 37.9] | 31.77 [25.0 to 40.3] | 39.02 [30.4 to 50.0] | 32.29 [25.3 to 41.2] | 32.99 [25.9 to 42.0] | 30.44 [23.6 to 39.2] | 32.49 [25.5 to 41.4]
  A/H1N1 Day 29 | 476.69 [351.4 to 646.6] | 495.34 [370.7 to 661.8] | 430.24 [322.8 to 573.4] | 596.45 [442.5 to 804.0] | 660.96 [493.1 to 886.0] | 634.42 [474.5 to 848.3] | 730.30 [538.8 to 989.8] | 465.89 [348.5 to 622.8]
  B/Yamagata Day 1 | 14.80 [12.8 to 17.2] | 15.53 [13.5 to 17.9] | 18.04 [15.7 to 20.8] | 18.01 [15.6 to 20.8] | 16.05 [13.9 to 18.5] | 15.84 [13.7 to 18.3] | 14.92 [12.9 to 17.3] | 14.63 [12.7 to 16.9]
  B/Yamagata Day 29 | 43.60 [37.6 to 50.5] | 43.1 [37.5 to 49.6] | 56.7 [49.4 to 65.1] | 54.23 [46.9 to 62.6] | 58.79 [51.0 to 67.7] | 51.38 [44.6 to 59.1] | 54.7 [47.2 to 63.4] | 52.65 [45.8 to 60.6]
  B/Victoria Day 1 | 35.10 [28.1 to 43.9] | 43.96 [35.5 to 54.4] | 38.15 [30.9 to 47.1] | 41.08 [33.0 to 51.1] | 39.86 [32.2 to 49.4] | 44.56 [36.0 to 55.1] | 38.07 [30.5 to 47.6] | 34.77 [28.1 to 43.0]
  B/Victoria Day 29 | 112.86 [93.4 to 136.3] | 117.97 [98.5 to 141.2] | 157.54 [131.8 to 188.3] | 168.62 [140.1 to 203.0] | 173.89 [144.9 to 208.6] | 152.41 [127.2 to 182.6] | 161.86 [134.0 to 195.5] | 146.56 [122.4 to 175.5]

10. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) (GMR is GMT Ratio of aQII Formulation/Licensed QII) for the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Microneutralization Assay
Time Frame: 28 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 105 | 106 | 99 | 102 | 104 | 95 | 104
Ratio
  A/H1N1 GMR (aQII/QII) | 1.04 [0.68 to 1.58] | 0.90 [0.59 to 1.37] | 1.25 [0.82 to 1.91] | 1.39 [0.91 to 2.11] | 1.33 [0.87 to 2.03] | 1.53 [1.00 to 2.35] | 0.98 [0.64 to 1.49]
  B/Yamagata GMR (aQII/QII) | 0.99 [0.81 to 1.21] | 1.30 [1.06 to 1.59] | 1.24 [1.01 to 1.53] | 1.35 [1.10 to 1.65] | 1.18 [0.96 to 1.44] | 1.25 [1.02 to 1.54] | 1.21 [0.99 to 1.48]
  B/Victoria GMR (aQII/QII) | 1.05 [0.81 to 1.36] | 1.40 [1.08 to 1.81] | 1.49 [1.15 to 1.94] | 1.54 [1.19 to 2.00] | 1.35 [1.04 to 1.75] | 1.43 [1.10 to 1.87] | 1.30 [1.00 to 1.68]

11. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving Seroconversion for the A/H1N1, B/Victoria and B/Yamagata Strains by MN Assay
Description: as for outcome 3
Time Frame: 28 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 95 | 105 | 106 | 99 | 102 | 104 | 95 | 104
percentage of subjects
  A/H1N1 Day 29 | 73.7 [63.6 to 82.2] | 82.9 [74.3 to 89.5] | 82.1 [73.4 to 88.8] | 79.8 [70.5 to 87.2] | 87.3 [79.2 to 93.0] | 83.7 [75.1 to 90.2] | 87.4 [79.0 to 93.3] | 87.5 [79.6 to 93.2]
  B/Yamagata Day 29 | 31.6 [22.4 to 41.9] | 27.6 [19.3 to 37.2] | 39.6 [30.3 to 49.6] | 38.4 [28.8 to 48.7] | 45.1 [35.2 to 55.3] | 37.5 [28.2 to 47.5] | 40.0 [30.1 to 50.6] | 42.3 [32.7 to 52.4]
  B/Victoria Day 29 | 37.9 [28.1 to 48.4] | 35.2 [26.2 to 45.2] | 48.1 [38.3 to 58.0] | 44.4 [34.5 to 54.8] | 50.0 [39.9 to 60.1] | 42.3 [32.7 to 52.4] | 45.3 [35.0 to 55.8] | 42.3 [32.7 to 52.4]

12. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) for the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Hemagglutination Inhibition (HI) Assay
Time Frame: 180 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 94 | 106 | 105 | 99 | 102 | 97 | 94 | 102
titer
  A/H1N1 Day 181 | 110.69 [89.3 to 137.2] | 95.07 [77.7 to 116.3] | 78.87 [64.4 to 96.5] | 86.67 [70.3 to 106.8] | 92.45 [75.3 to 113.5] | 78.23 [63.4 to 96.6] | 85.50 [69.0 to 105.9] | 86.67 [70.6 to 106.5]
  B/Yamagata Day 181 | 25.05 [21.3 to 29.5] | 26.58 [22.8 to 31.0] | 26.71 [22.9 to 31.2] | 24.89 [21.2 to 29.2] | 25.52 [21.8 to 29.8] | 24.73 [21.1 to 29.0] | 27.00 [22.9 to 31.8] | 27.33 [23.4 to 32.0]
  B/Victoria Day 181 | 55.42 [44.5 to 69.1] | 53.30 [43.3 to 65.6] | 59.26 [48.2 to 72.9] | 56.00 [45.2 to 69.4] | 56.97 [46.1 to 70.4] | 55.86 [45.0 to 69.3] | 68.07 [54.6 to 84.8] | 57.94 [46.9 to 71.5]

13. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) (GMR is GMT Ratio of aQII Formulation/Licensed QII) for the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Hemagglutination Inhibition (HI) Assay
Time Frame: 180 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 106 | 105 | 99 | 102 | 97 | 94 | 102
Ratio
  A/H1N1 Day 181 (aQII/QII) | 0.86 [0.64 to 1.15] | 0.71 [0.53 to 0.96] | 0.78 [0.58 to 1.05] | 0.84 [0.62 to 1.12] | 0.71 [0.52 to 0.95] | 0.77 [0.57 to 1.04] | 0.78 [0.58 to 1.05]
  B/Yamagata Day 181 (aQII/QII) | 1.06 [0.85 to 1.33] | 1.07 [0.85 to 1.34] | 0.99 [0.79 to 1.25] | 1.02 [0.81 to 1.28] | 0.99 [0.79 to 1.24] | 1.08 [0.86 to 1.36] | 1.09 [0.87 to 1.37]
  B/Victoria Day 181 (aQII/QII) | 0.96 [0.71 to 1.30] | 1.07 [0.79 to 1.45] | 1.01 [0.74 to 1.37] | 1.03 [0.76 to 1.39] | 1.01 [0.74 to 1.37] | 1.23 [0.90 to 1.68] | 1.05 [0.77 to 1.42]

14. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects With HI Titer ≥1:40 for A/H1N1, B/Yamagata and B/Victoria Strains (HI Assay)
Time Frame: 180 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 94 | 106 | 105 | 99 | 102 | 97 | 94 | 102
percentage
  A/H1N1 Day 181 | 87.2 [78.8 to 93.2] | 85.8 [77.7 to 91.9] | 80.0 [71.1 to 87.2] | 82.8 [73.9 to 89.7] | 87.3 [79.2 to 93.0] | 80.4 [71.1 to 87.8] | 83.0 [73.8 to 89.9] | 81.4 [72.4 to 88.4]
  B/Yamagata Day 181 | 42.6 [32.4 to 53.2] | 42.5 [32.9 to 52.4] | 49.5 [39.6 to 59.5] | 44.4 [34.5 to 54.8] | 40.2 [30.6 to 50.4] | 40.2 [30.4 to 50.7] | 44.7 [34.4 to 55.3] | 44.1 [34.3 to 54.3]
  B/Victoria Day 181 | 71.3 [61.0 to 80.1] | 75.5 [66.2 to 83.3] | 74.3 [64.8 to 82.3] | 71.7 [61.8 to 80.3] | 72.5 [62.8 to 80.9] | 74.2 [64.3 to 82.6] | 73.4 [63.3 to 82.0] | 71.6 [61.8 to 80.1]

15. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) for the A/H1N1, A/H3N2, B/Victoria and B/Yamagata Vaccine Strains by MN Assay
Time Frame: 180 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 94 | 106 | 105 | 99 | 102 | 97 | 94 | 102
titer
  A/H1N1 Day 181 | 516.06 [382.5 to 696.2] | 529.64 [399.8 to 701.7] | 427.95 [322.9 to 567.2] | 615.44 [459.8 to 823.7] | 562.64 [422.6 to 749.1] | 518.67 [386.8 to 695.5] | 644.81 [478.4 to 869.0] | 493.66 [370.8 to 657.3]
  A/H3N2 Day 181 | 73.72 [60.7 to 89.5] | 70.50 [58.7 to 84.6] | 74.71 [62.2 to 89.7] | 91.77 [76.0 to 110.9] | 83.3 [69.2 to 100.3] | 85.11 [70.4 to 103.0] | 90.00 [74.2 to 109.2] | 63.44 [52.7 to 76.4]
  B/Yamagata Day 181 | 26.19 [22.8 to 30.1] | 26.38 [23.1 to 30.1] | 28.53 [25.0 to 32.5] | 31.48 [27.5 to 36.1] | 31.3 [27.4 to 35.8] | 27.82 [24.3 to 31.9] | 30.96 [26.9 to 35.6] | 32.20 [28.2 to 36.8]
  B/Victoria Day 181 | 175.30 [146.4 to 209.9] | 180.26 [152.1 to 213.6] | 209.57 [176.8 to 248.4] | 246.04 [206.4 to 293.3] | 238.56 [200.7 to 283.6] | 199.67 [167.3 to 238.4] | 286.95 [239.7 to 343.5] | 218.44 [183.8 to 259.6]

16. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) (GMR is GMT Ratio of aQII Formulation/Licensed QII) for the A/H1N1, A/H3N2, B/Victoria and B/Yamagata Vaccine Strains by MN Assay
Time Frame: 180 days post-vaccination
Population: The analysis population is PPS Immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
Number analyzed (Participants) | 106 | 105 | 99 | 102 | 97 | 94 | 102
Ratio
  A/H1N1 Day 181 (aQII/QII) | 1.03 [0.68 to 1.55] | 0.83 [0.55 to 1.25] | 1.19 [0.79 to 1.81] | 1.09 [0.72 to 1.65] | 1.01 [0.66 to 1.53] | 1.25 [0.82 to 1.90] | 0.96 [0.63 to 1.45]
  A/H3N2 Day 181 (aQII/QII) | 0.96 [0.73 to 1.25] | 1.01 [0.78 to 1.32] | 1.24 [0.95 to 1.63] | 1.13 [0.86 to 1.48] | 1.15 [0.88 to 1.51] | 1.22 [0.93 to 1.60] | 0.86 [0.66 to 1.13]
  B/Yamagata Day 181 (aQII/QII) | 1.01 [0.83 to 1.22] | 1.09 [0.90 to 1.32] | 1.20 [0.99 to 1.46] | 1.19 [0.99 to 1.45] | 1.06 [0.87 to 1.29] | 1.18 [0.97 to 1.44] | 1.23 [1.01 to 1.49]
  B/Victoria Day 181 (aQII/QII) | 1.03 [0.80 to 1.32] | 1.20 [0.93 to 1.53] | 1.40 [1.09 to 1.80] | 1.36 [1.06 to 1.75] | 1.14 [0.89 to 1.47] | 1.64 [1.27 to 2.11] | 1.25 [0.97 to 1.60]

ADVERSE EVENTS:
Time Frame: Time frame for all-cause mortality: 6 months SAEs: Day 1 to Day 181, Nonserious unsolicited AEs: Day 1 to Day 29, Solicited AEs: Day 1 to Day 7 after vaccination
Description: SAEs, nonserious unsolicited AEs, and solicited AEs are reported in this Adverse Events section
Arm/Group | Group H Licensed QII Active Comparator | Group A aQII-1 Investigational | Group E aQII-9 Investigational | Group C aQII-6 Investigational | Group F aQII-10 Investigational | Group B aQII-3 Investigational | Group D aQII-7 Investigational | Group G aQII-11 Investigational
All-Cause Mortality (participants affected / at risk) | 1/97 | 0/107 | 0/108 | 0/103 | 1/106 | 1/107 | 1/101 | 0/109
Serious Adverse Events (participants affected / at risk) | 8/97 | 1/107 | 1/108 | 3/103 | 5/106 | 3/107 | 2/101 | 2/109
Other Adverse Events (participants affected / at risk) | 55/97 | 74/107 | 80/108 | 79/103 | 91/106 | 81/107 | 72/101 | 89/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group H Licensed QII Active Comparator (N=97) | Group A aQII-1 Investigational (N=107) | Group E aQII-9 Investigational (N=108) | Group C aQII-6 Investigational (N=103) | Group F aQII-10 Investigational (N=106) | Group B aQII-3 Investigational (N=107) | Group D aQII-7 Investigational (N=101) | Group G aQII-11 Investigational (N=109)
retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group H Licensed QII Active Comparator (N=97) | Group A aQII-1 Investigational (N=107) | Group E aQII-9 Investigational (N=108) | Group C aQII-6 Investigational (N=103) | Group F aQII-10 Investigational (N=106) | Group B aQII-3 Investigational (N=107) | Group D aQII-7 Investigational (N=101) | Group G aQII-11 Investigational (N=109)
nausea (Gastrointestinal disorders) | 7 (7) | 8 (8) | 10 (10) | 12 (12) | 19 (20) | 9 (9) | 10 (10) | 16 (17)
chills (General disorders) | 8 (8) | 6 (6) | 9 (9) | 10 (11) | 18 (19) | 10 (10) | 13 (13) | 20 (21)
fatigue (General disorders) | 25 (27) | 25 (25) | 34 (36) | 36 (37) | 41 (42) | 27 (29) | 31 (31) | 47 (48)
induration (General disorders) | 1 (1) | 9 (9) | 10 (10) | 7 (7) | 14 (14) | 9 (9) | 10 (10) | 15 (15)
injection site pain (General disorders) | 29 (29) | 53 (53) | 61 (61) | 66 (66) | 70 (70) | 53 (53) | 53 (53) | 71 (71)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 8 (8) | 4 (4) | 4 (4) | 6 (6) | 5 (5) | 5 (5) | 4 (4)
loss of appetite (Metabolism and nutrition disorders) | 4 (4) | 11 (11) | 8 (8) | 14 (14) | 14 (14) | 6 (6) | 9 (9) | 21 (21)
arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 19 (20) | 19 (19) | 21 (21) | 33 (34) | 25 (28) | 22 (24) | 25 (27)
myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 16 (16) | 20 (20) | 24 (24) | 34 (35) | 24 (25) | 19 (19) | 27 (27)
headache (Nervous system disorders) | 18 (18) | 27 (27) | 28 (28) | 30 (31) | 42 (43) | 31 (32) | 29 (29) | 39 (41)
erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 9 (9) | 7 (7) | 12 (12) | 10 (10) | 9 (9) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT04782323/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT04782323/SAP_001.pdf